CLINICAL TRIAL: NCT06923345
Title: Modified Long-Course Radiotherapy (Reduced vs. Conventional CTV), Sequential Chemotherapy and PD-1 Inhibitor in Locally Advanced, MSS, Mid-Low Rectal Cancer: An Open-Label, Two-Arm, Randomized, Prospective Phase II Clinical Trial (MODIFI-RC-I)
Brief Title: Modified Long-Course Radiotherapy Followed by Chemotherapy and PD-1 Inhibitor for MSS/pMMR High-risk Mid/Low LARC (MODIFI-RC-I)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Assistant President of the Sixth Affiliated Hospital of Sun Yat-sen University; Chief Physician of Department of Colorectal Surgery, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-147
Record Dates: First submitted 2025-04-01; First posted 2025-04-11 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer; Neoadjuvant Therapies; Immune Checkpoint Therapy; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Select-a-winner design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced CTV (Experimental): Patients will receive long-course radiotherapy with selective reduced CTV irradiation, concurrently with 3 cycles of CAPOX chemotherapy and PD-1 inhibitor. After radiotherapy, they will receive an additional 3 cycles of CAPOX chemotherapy and PD-1 inhibitor, followed by either total mesorectal excision (TME) surgery or watch-and-wait observation.
  Interventions: Combination Product: Reduced CTV
- Conventional CTV (Experimental): Patients will receive long-course radiotherapy with conventional CTV irradiation, concurrently with 3 cycles of CAPOX chemotherapy and PD-1 inhibitor. After radiotherapy, they will receive an additional 3 cycles of CAPOX chemotherapy and PD-1 inhibitor, followed by either total mesorectal excision (TME) surgery or watch-and-wait observation.
  Interventions: Combination Product: Conventional CTV

INTERVENTIONS:
Combination Product: Reduced CTV — Long-course radiotherapy with selective CTV reduction (lower to S2/S3 level) + CAPOX + PD-1 inhibitor.
  After treatment, patients will undergo TME surgery or a watch-and-wait approach, depending on response.
  Arms: Reduced CTV
Combination Product: Conventional CTV — Long-course radiotherapy with conventional CTV irradiation + CAPOX + PD-1 inhibitor.
  After treatment, patients will undergo TME surgery or a watch-and-wait approach, depending on response.
  Arms: Conventional CTV

SUMMARY:
The goal of this clinical trial is to evaluate whether a total neoadjuvant therapy (TNT) regimen combining long-course chemoradiotherapy, sequential chemotherapy, and PD-1 inhibitor can improve response rates, enhance tolerability, and improve prognosis in patients with locally advanced, microsatellite-stable (MSS) rectal cancer.

The main questions it aims to answer are:

Does this TNT approach improve complete response (CR) rates?

How does selective reduction of clinical target volume (CTV) to S2/S3 level compare with conventional CTV irradiation in terms of efficacy and safety?

Researchers will compare a selective CTV reduction group and a conventional CTV irradiation group to assess differences in treatment outcomes, including complete response, tumor regression grading (TRG), organ preservation, R0 resection rates, and long-term survival.

Participants will:

Receive long-course chemoradiotherapy with either conventional or reduced CTV irradiation.

Undergo sequential chemotherapy.

Receive PD-1 inhibitor treatment.

Be monitored for safety, tumor regression, and long-term survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signs a written informed consent form.
* Aged between 18 and 75 years at enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival of more than 2 years.
* Histologically confirmed rectal adenocarcinoma.
* Tumor biopsy immunohistochemistry indicating pMMR (MSH1, MSH2, MSH6, and PMS2 all positive) or genetic testing confirming MSS.
* According to the 8th edition of the AJCC TNM classification, high-resolution MRI ± endorectal ultrasound confirms clinical staging as cT3-4NanyM0 or cTxN+M0 (stage II-III rectal cancer). MRI confirms the tumor is located below the peritoneal reflection without lateral lymph node metastasis.
* Before study enrollment, a responsible surgical attending physician must evaluate the patient's medical history to confirm eligibility for R0 resection with curative intent.
* No prior systemic or local anti-tumor treatment for rectal cancer, including radiotherapy, chemotherapy, immunotherapy, biologics, or small-molecule targeted therapy.
* Willing to provide tumor tissue and peripheral blood samples for research purposes during screening and throughout the study.
* Adequate organ function:
* Hematology (without recent blood transfusions or growth factor support within 7 days before treatment):

  * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L (1,500/mm³)
  * Platelet count ≥ 100 × 10⁹/L (100,000/mm³)
  * Hemoglobin ≥ 90 g/L
* Renal function:

  * Estimated creatinine clearance (CrCl) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)
  * Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g
* Liver function:

  * Total bilirubin (TBil) ≤ 1.5 × upper limit of normal (ULN)
  * AST and ALT ≤ 2.5 × ULN
  * Serum albumin (ALB) ≥ 28 g/L
* Coagulation function:

  o INR and APTT ≤ 1.5 × ULN
* Cardiac function:

  o Left ventricular ejection fraction (LVEF) ≥ 50%
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 3 days before starting study treatment. If a urine pregnancy test result is unclear, a confirmatory serum pregnancy test must be conducted. Participants with childbearing potential who engage in sexual activity with non-sterilized male partners must use highly effective contraception from screening until 120 days after the last dose of study treatment. The use of periodic abstinence and fertility awareness methods is not considered acceptable contraception.
* Definition of females of childbearing potential (FCBP): Women who have not undergone surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or total hysterectomy) or who have not been naturally postmenopausal for at least 12 consecutive months (confirmed by FSH levels within the postmenopausal range).
* Highly effective contraception methods: Must have a failure rate of <1% per year when used consistently and correctly. In addition to barrier methods, FCBP must use an additional hormonal contraceptive method (e.g., oral contraceptives).
* Participants must be willing and able to comply with study visit schedules, treatment plans, laboratory tests, and other study-related requirements.

Exclusion Criteria:

* Presence of suspected metastatic lesions or locally advanced unresectable disease, regardless of disease stage.
* Diagnosis of other malignancies within the past five years, except for patients with malignancies cured through local treatment (e.g., basal or squamous cell skin cancer, superficial bladder cancer, ductal carcinoma in situ of the breast).
* Concurrent enrollment in another clinical study, unless it is an observational, non-interventional study or a follow-up phase of an interventional study.
* Presence of intestinal obstruction, perforation, or bleeding requiring emergency surgery.
* Multiple primary rectal cancers.
* History of pelvic or abdominal radiotherapy.
* Inability to swallow tablets, malabsorption syndrome, or any condition affecting gastrointestinal absorption.
* Prior systemic or local anti-tumor treatment for locally advanced rectal cancer, including radical surgery, chemotherapy, radiotherapy, immunotherapy (e.g., immune checkpoint inhibitors, immune cell therapy), biological agents, or targeted therapy.
* Use of nonspecific immunomodulatory treatment (e.g., interleukins, interferons, thymosin, TNF) within two weeks before study treatment (excluding IL-11 for thrombocytopenia); use of traditional Chinese medicine with anti-tumor indications within one week before study treatment.
* Active autoimmune disease requiring systemic treatment in the past two years, except for replacement therapy (e.g., thyroid hormone, insulin, corticosteroids for adrenal/pituitary insufficiency).
* History of non-infectious pneumonitis requiring systemic glucocorticoid therapy or interstitial lung disease.
* History of severe bleeding tendency, coagulopathy, or long-term anticoagulation therapy (e.g., atrial fibrillation with CHADS2 score ≥2).
* Uncontrolled comorbidities, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease, or psychiatric/social conditions limiting compliance.
* History of myocarditis, cardiomyopathy, malignant arrhythmias; hospitalization for unstable angina, congestive heart failure, or vascular diseases (e.g., aortic aneurysm requiring surgery) within 12 months before study treatment.
* History of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, chronic diarrhea).
* Severe infection within four weeks before study treatment, including sepsis or severe pneumonia requiring hospitalization; active infection requiring systemic therapy within ten days before study treatment (excluding antiviral therapy for HBV or HCV).
* Major surgery or severe trauma within 30 days before study treatment; minor surgery (excluding peripheral venous catheterization) within three days before study treatment.
* Immunodeficiency history, positive HIV test, or long-term use of systemic corticosteroids or immunosuppressants.
* Active tuberculosis or suspected TB requiring clinical exclusion; known active syphilis infection.
* History of allogeneic organ or hematopoietic stem cell transplantation.
* Untreated active HBV infection (HBsAg-positive with HBV-DNA > 1000 copies/ml or 200 IU/ml); active HCV infection (HCV antibody-positive with detectable HCV-RNA).
* Live vaccine administration within 30 days before study treatment or planned during the study period.
* Known hypersensitivity to any study drug component or history of severe hypersensitivity reactions to monoclonal antibodies.
* History of psychiatric disorders, substance abuse, alcohol dependence, or drug addiction.
* Pregnant or breastfeeding women.
* Any disease, treatment, or laboratory abnormality that may confound study results, interfere with full study participation, or is not in the participant's best interest.
* Non-malignant or tumor-related systemic diseases or symptoms causing high medical risk or uncertainty in survival assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | From enrollment to 2 weeks after finishing TNT
  Evaluate whether total neoadjuvant therapy (TNT) with long-course chemoradiotherapy (selective vs. conventional CTV), sequential CAPOX chemotherapy, and PD-1 inhibitor improves the complete response (CR) rate in locally advanced MSS rectal cancer.

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | From enrollment to 2 weeks after finishing TNT
Tumor downstaging rate | From enrollment to 2 weeks after finishing TNT
Watch-and-wait rate | From enrollment to 2 weeks after finishing TNT
Sphincter preservation rate | From date of randomization until the date of surgery or the date of watch-and-wait for CR patients
R0 resection rate | From date of randomization until the date of surgery or the date of watch-and-wait for CR patients
3-year event-free survival (EFS) rate | From enrollment to 3 years after finishing Surgery
3-year distant metastasis rate | From enrollment to 3 years after finishing Surgery
3-year local recurrence rate | From enrollment to 3 years after finishing Surgery
3-year overall survival (OS) rate | From enrollment to 3 years after finishing Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No